CLINICAL TRIAL: NCT06616285
Title: The Effects of a Hungarian Multidomain Lifestyle Intervention on Brain Health in Older Adults
Acronym: HUN-MLI-BRAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Research Centre for Natural Sciences (Other)
Collaborators: HUN-REN Institute of Experimental Medicine (Unknown); Semmelweis University (Other)
Responsible Party: Principal Investigator, Vidnyánszky Zoltán, Director of Brain Imaging Centre, HUN-REN Centre for Natural Sciences, Research Centre for Natural Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 298/2/2023/HF
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-09

CONDITIONS: Neurocognitive Aging; Healthy Aging
Keywords: Brain; Healthy Aging; Multidomain intervention; Neurocognitive Aging

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. Participants will be randomised either into the Folk Dance Multidomain Lifestyle Intervention Group or the Self-Guided Multidomain Lifestyle Intervention Group. The intervention will be delivered over a period of 6 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Baseline assessments will be conducted at the research centre prior to randomisation. After baseline assessments and randomisation, two members of the research team will be unblinded to group allocation in order to coordinate the intervention. Post-intervention measurements and data analyses will be conducted by researchers and trained research assistants who are blind to participant randomisation and are not present during the intervention sessions. Participants will be instructed not to disclose their randomisation status during any of the assessment sessions or in-house visits. Participants and intervention staff will be aware of their group allocation. The intervention staff will not conduct any assessment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folk Dance Multidomain Lifestyle Intervention (Active Comparator): Participants will receive structured, intensive lifestyle intervention through group and individual sessions. Main lifestyle components included: diet, physical exercise, mental stimulation, cardiovascular/metabolic risk monitoring, social interaction. The intervention will last for 6 months.
  Interventions: Behavioral: Folk Dance Multidomain Lifestyle Intervention
- Self-Guided Multidomain Lifestyle Intervention (Sham Comparator): Participants will receive multi-domain lifestyle intervention that provides guidance on healthy diet, physical activity, and mental stimulation, and cardiovascular/metabolic risk factors monitoring. The intervention will last for 6 months.
  Interventions: Behavioral: Self-Guided Multidomain Lifestyle Intervention

INTERVENTIONS:
Behavioral: Self-Guided Multidomain Lifestyle Intervention — Participants will receive guidance on healthy dietary habits, physical activity, mental stimulation, and cardiovascular/metabolic monitoring based on national recommendations and individual consultations with the study physician. Based on this guidance, participants will create their own healthy lifestyle plan. Participants' cardiovascular/metabolic risk factors will be regularly monitored.
  Arms: Self-Guided Multidomain Lifestyle Intervention
Behavioral: Folk Dance Multidomain Lifestyle Intervention — Participants will receive structured, intensive lifestyle intervention with the following components: diet, physical exercise, mental stimulation, cardiovascular/metabolic risk monitoring, social interaction.
  One-hour long folk dancing sessions, delivered by professional teachers 3 times weekly, will provide opportunities for physical and mental exercise and social interaction. These sessions were specifically developed to foster physical and mental stimulation through the learning of coordinated movement and different choreographies (rhythmic and gradually more complex movements with folk songs) individually, in pairs, and circles. As such, social stimulation is naturally embedded in the sessions.
  Participants will receive advice about diet and cardiovascular/metabolic risk factors based on national recommendations via group sessions and individual consultations. Participants' cardiovascular/metabolic risk factors will be regularly monitored.
  Arms: Folk Dance Multidomain Lifestyle Intervention

SUMMARY:
Maintaining brain health in older adults is a critical social and economic challenge given the rising prevalence of neurodegenerative disorders. Despite extensive research, effective pharmacological treatments for dementia remain limited, emphasising the need for early diagnosis and prevention of cognitive decline. Research suggests that lifestyle and modifiable factors account for approximately 40% of dementia risk, highlighting the potential of personalised lifestyle interventions to delay or prevent the onset of dementia. The original FINGER study demonstrated that a multi-domain lifestyle intervention simultaneously targeting dietary habits, physical and cognitive activity, as well as social interactions can effectively prevent cognitive decline and dementia.

The HUN-MLI-BRAIN trial investigates the impact of a Hungarian lifestyle intervention on brain health in older adults and is based on the FINGER multi-domain intervention. This randomised controlled study aims to maintain and enhance neurocognitive function and prevent cognitive decline in older adults through a multi-domain lifestyle program, which simultaneously targets dietary habits, physical and cognitive activity, and social engagement.

The primary goal of the HUN-MLI-BRAIN trial is to evaluate the impact of the intervention programme on neurocognitive functions and adaptive changes in large-scale brain networks at the individual level using the precision structural and functional MRI methods as well as resting-state EEG frequency-domain analyses. In addition, the influence of the intervention will be assessed in a wide range of cognitive and personal domains. The potential relationship between brain structure and function, cognitive performance, lifestyle factors, and dementia risk factors will be evaluated.

80 people without substantial cognitive impairment or dementia will be recruited into the programme in Budapest, Hungary. Participants will be randomly allocated 1:1 either to the multi-domain, folk dancing lifestyle intervention group or the self-guided, multi-domain lifestyle intervention group. The self-guided intervention encompasses multi-domain lifestyle recommendations on diet, physical and mental training, and health checks via the Polar Pacer smart watch. The folk dancing intervention includes structured, one-hour folk dancing sessions three times per week, which were specifically developed to foster physical and cognitive function whilst facilitating social interaction. Participants in this group will also receive intensive and tailored lifestyle recommendations aimed at improving physical and mental functioning. The duration of the intervention programme is 6 months. Participants will complete assessment visits before and after the intervention.

The HUN-MLI-BRAIN trial holds significant potential for advancing our understanding of how lifestyle interventions may impact brain function. The use of advanced, precision neuroimaging techniques will offer novel insights into the adaptive changes in brain networks and potentially lead to more effective, personalised interventions for maintaining brain health in older adults.

DETAILED DESCRIPTION:
Participants will first complete a short phone call designed to screen for eligibility and exclusion criteria. Selected participants will be invited for an in-house assessment, during which they will be further screened for cognitive, physical, and lifestyle risk factors as well as MRI scanning compatibility. Using the Mini-Mental State Examination, a board-certified neurologist will also screen participants for cognitive impairment.

Participants will be invited for several baseline and post-intervention assessments on separate days. First, eligible participants will complete a complex cognitive assessment. Next, EEG and pupillometry data will be collected from participants during rest and the completion of a probabilistic reversal learning task, which evaluates reinforcement learning behaviour and related neural mechanisms. Crucially, participants will also complete structural and functional MRI assessments. Using precision resting-state functional MRI, the study will examine large-scale brain network segregation as well as network-specific within and cross-network connectivity changes, which are known to be affected by ageing and neuropsychiatric diseases. A novel multi-echo multiband sequence, with enhanced BOLD signal sensitivity and reduced image artefacts, will be employed to improve test-retest reliability. During data collection, special care will be taken to ensure the availability of a sufficient amount of clean resting-state fMRI data, which is essential to ensure the accuracy and validity of the findings. Finally, blood samples will be collected from each participant.

Following all baseline assessments, participants will be randomised into the folk dancing or self-guided lifestyle intervention groups. Block-randomisation will be computerised with a targeted assignment ratio of 1:1 and stratification for age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65-75 years
* Proficiency in the local (Hungarian) language
* Ability to perform all the three components of the Short Physical Performance Battery (score of at least 1 in each component)

Exclusion Criteria:

* Previous diagnosis of mild cognitive impairment or dementia, including current use of medications for memory impairment
* Suspected mild cognitive impairment or dementia after screening assessments, based on clinical judgement
* Contraindication for MRI scanning (e.g., metal implants, claustrophobia, excessive movement, etc.)
* History of any significant neurological condition, including Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumours, progressive supranuclear palsy, seizure disorder, subdural heamatoma, multiple sclerosis, or history of stroke, transient ischemic attack, or any significant head trauma with persistent neurologic sequelae or known structural brain abnormalities
* History of major depression, bipolar disorder, schizophrenia
* Chronic medication use that could reasonably affect cognition, movement, or brain imaging measures
* Active substance-related and addictive disorders
* Current use of narcotics and psychoactive medications
* Cognitive impairment based on the Mini-Mental State Examination (MMSE, raw score less than 26)
* Reduced capacity for decision-making, unable to provide consent or complete study assessments, based on clinical judgement
* Conditions that prevent safe study participation
* Current significant medical problems (e.g., malignant disease, cardiovascular disease, conduction disorder)
* History within the last 2 years of treatment for primary or recurrent malignant disease
* Poorly controlled or uncontrolled diabetes mellitus, cardiovascular, conduction, or pulmonary disease
* Conditions that prevent cooperation: severe visual, auditory, or communication impairment (i.e., colour blindness, uncorrected hearing loss)
* PI/Study Clinician discretion regarding medical status, suitability of participation, or concerns about adherence to intervention
* Ongoing participation in another clinical intervention study

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Brain Functional Connectivity Measured with Resting-State fMRI | Baseline, 6 month
  Multi-echo functional MRI (3T Siemens Prisma scanner) measure of individual large-scale brain network segregation as well as network-specific within and cross-network connectivity changes will be derived. Network segregation will be estimated by computing the difference between within-network connectivity and between-network connectivity, normalised by the total connectivity.
Changes in Brain Function Measured with Resting-State EEG | Baseline, 6 month
  Resting-state neural activity will be recorded via a 64-channel Brain Products actiCAP EEG device.
  Individual-level periodic and aperiodic α peak frequency will be computed.

SECONDARY OUTCOMES:
Connectivity Changes in Brain Reward System | Baseline, 6 month
  Cortical and subcortical resting-state multi-echo fMRI effective connectivity of brain regions associated with reward and motivation will be estimated using dynamic causal modelling.
Connectivity Changes in the Brain's Default Mode Network | Baseline, 6 month
  Cortical and subcortical resting-state multi-echo fMRI effective connectivity of the default mode network will be estimated using dynamic causal modelling.
Changes in Hippocampal Volume | Baseline, 6 month
  The volumes of the hippocampal subfields will be computed using proton density-weighted MRI.
Changes in the Striatal Volume | Baseline, 6 month
  The volumes of the striatal nuclei will be derived from T1 weighted MRI.
Changes in the Volume of Neuromodulatory Nuclei | Baseline, 6 month
  The integrity of the substantia nigra-ventral tegmental area (SN-VTA) and locus coeruleus (LC) will be computed based on magnetization transfer-weighted MRI.
Changes in Brain Age | Baseline, 6 month
  Individual brain age will be estimated using T1-weighted MRI images utilising pre-trained deep neural networks specifically trained for brain age prediction.
Changes Resting-State EEG Frequency Band Ratio Measures | Baseline, 6 month
  The relative contribution of resting-state EEG frequency band measures will be computed (alpha, beta, delta, theta frequency bands).
Changes in Feedback-Related EEG and Pupil Responses | Baseline, 6 month
  Changes in feedback-related EEG (early and late feedback components, P300 and Error-related Negativity ERPs) and pupil responses will be measured during the Probabilistic Reversal Learning Task. During this task, participants have to choose between two abstract symbols. In the reward condition, participants receive positive (reward, +1 point) and neutral (zero point) feedback. In the punishment conditions, participants receive negative (punishment, -1 point) or neutral feedback. Participants complete 2 blocks of 80 trials of each condition (a total of 320 trials). In any given trial, one symbol is associated with a high (80%) and the other with a low (20%) probability of reward or lack of punishment. A reversal in reward contingencies is introduced 3-7 times per block. Participants are instructed to maximise the number of points earned throughout the experiment and are financially compensated based on their performance in the task.
Changes in Subjective Cost of Cognitive Effort | Baseline, 6 month
  Changes in the subjective cost of cognitive effort will be measured using the Cognitive Effort Discounting Paradigm.
Changes in Global Cognitive Function | Baseline, 6 month
  Global cognitive function will be assessed using a composite score, which will be derived from a series of neuropsychological tests, including Verbal Episodic Memory Test, Location Learning Test, Digit Span, Verbal Fluency, Trail-Making Test, Victoria Stroop Test, and Digit Symbol Substitution Test. Scores from each test will be transformed into z-scores and then averaged to create a composite score. Higher scores indicate better performance.
Changes in Episodic Memory | Baseline, 6 month
  Episodic Memory will be a composite score obtained from the Verbal Episodic Memory Test and the Location Learning Test. The Episodic Memory composite is calculated in the same way as the composite score for global cognitive function.
Changes in Executive Function | Baseline, 6 month
  Executive Function will be a composite score obtained from Digit Span, Digit Symbol Substitution, Trail Making Test Part B, Victoria Stroop Test, and Verbal Fluency. The Executive Function composite is calculated in the same way as the composite score for global cognitive function.
Changes in Processing Speed | Baseline, 6 month
  Processing Speed will be a composite score obtained from Digit Symbol Substitution and Trail Making Test Part A. The Processing Speed composite is calculated in the same way as the composite score for global cognitive function.
Changes in Blood Biomarkers | Baseline, 6 month
  Inflammatory cytokines, C-reactive protein, glial fibrillary acidic protein, Clustering, Brain Derived Neurotrophic factor, Insulin Growth Factor-1
Changes in Anthropometry | Baseline, 6 month
  Waist circumference (cm) will be measured.
Changes in Body Mass Index (BMI) | Baseline, 6 month
  Body Mass Index (BMI) is a measure of body fat based on height and weight for adult men and women. BMI will be expressed in kg/m^2.
Changes in Systolic Blood Pressure | Baseline, 6 month
  Systolic blood pressure (mmHg) will be recorded using calibrated blood pressure monitors.
Changes in Diastolic Blood Pressure | Baseline, 6 month
  Diastolic blood pressure (mmHg) will be recorded using calibrated blood pressure monitors.
Changes in Hand Grip Strength | Baseline, 6 month
  Hand grip strength will be quantified using a hand dynamometer, with higher values indicating greater muscle strength.
Changes in Physical Performance | Baseline, 6 month
  Physical performance will be assessed using the Short Physical Performance Battery (SPPB), which assesses balance, mobility, and muscle strength in older adults. The total score is the sum of the three components and ranges between 0 and 12, with higher scores indicating a better outcome. Only individuals with a score ≥ 1 in each subtest will be included in the study.
Changes in Physical Activity - Self-reported | Baseline, 6 month
  Subjective physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ). It measures the types of PA intensity and time spent sitting that individuals do as part of their daily lives. Total subjective PA will be assessed in MET-min/week and time spent sitting will be assessed in min/day.
Changes in Physical Activity | 7-day wear period every 2 months
  Changes in physical activity will be objectively measured using the Polar Pacer smart watch. Participants will be asked to wear the watch for 7 consecutive days every 2 months during the intervention. The device will track participants' heart rate, heart rate variability (calculated from pulse lengths), and MET (Metabolic Equivalent of Task).
Changes in Sleep | 7-day wear period every 2 months
  Sleep will be tracked via the Polar Pacer smart watch. Participants will be asked to wear the watch for 7 consecutive days every 2 months during the intervention. The device will monitor participant's total sleep duration, the time spent in REM sleep, deep sleep, and light sleep as well as the percentage of each of the three sleep stages compared to total sleep time. The watch will also estimate the amount of interrupted sleep and a total sleep score per night (ranging from 1 to 100).
Changes in Subjective Sleep Quality | Baseline, 6 month
  Subjective sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI). The global score ranges from 0 to 21, with higher scores indicating worse sleep quality.
Changes in Sleep Disorder | Baseline, 6 month
  The Athens Insomnia Scale (AIS) will be employed to assess the severity of insomnia. The total score ranges between 0 and 24, with higher scores indicating a more severe sleep disorder.
Changes in Depressive Symptoms | Baseline, 6 month
  Depressive symptoms will be evaluated using the Geriatric Depression Scale (GDS) and the Patient Health Questionnaire (PHQ-9). The GDS score ranges from 0 to 15, while the PHQ-9 provides a severity score ranging from 0 to 27. A score of ≥ 5 on either scale is indicative of the presence of depressive symptoms.
Changes in Well-Being | Baseline, 6 month
  Well-being will be measured using the Hungarian version of the WHO Well-Being Questionnaire (WBI-5). The score can range from 0 to 15 points. A higher score indicates a greater degree of positive psychological well-being.
Changes in Social Support | Baseline, 6 month
  Perceived social support of the individual from the family, friends, and significant others will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS). The total score on the MSPSS ranges from 10 to 50, with higher scores indicating greater perceived social support.
Changes in Lifestyle | Baseline, 6 month
  A self-reported lifestyle questionnaire will be completed, collecting information about social life, mental activities, eating habits, subjective memory, and health status.
Changes in Sarcopenia Symptoms | Baseline, 6 month
  The SARC-F questionnaire will be employed as a screening tool for sarcopenia. The scores range from 0 to 10, with a cutoff of ≥ 4, indicating the presence of sarcopenia.
Dementia Risk Score (CAIDE) | Baseline, 6 month
  Weighted sum of the following dementia risk factors: age, sex, educational level in years, total cholesterol, physical activity status, systolic blood pressure, BMI, and diabetes. Higher scores indicate an increased risk for dementia.

OTHER OUTCOMES:
Demographics and medical history | Baseline
  Individuals will be asked to provide information about their sociodemographic (age, sex, ethnicity), education, and employment status, as well as their family (dementia) and medical history (head injury, diabetes, sleep apnoea, cardiovascular diseases, COVID-19 history and vaccination), medication and substance use (smoking, alcohol).
Instrumental Activities of Daily Living (IADL) | Baseline
  The Lawton IADL will be used to assess the individual's functional ability to perform daily tasks such as shopping, preparing meals, taking medication, and managing finances. Scores range from 0 to 8, with higher scores indicating better performance, i.e., more independent functionality.
Dementia screening | Baseline
  The Mini-Mental State Examination (MMSE) will be used as a rapid screening instrument for dementia. It measures multiple cognitive domains, such as orientation, memory, attention and calculation, executive functions, visuospatial skills, abstraction. The scores range between 0 and 30, with the score of less than 26 indicating cognitive impairment. Participants who score below this cutoff will be excluded from this study.

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Vidnyánszky, Ph.D., DSc., Principal Investigator — HUN-REN Centre for Natural Sciences
Locations (1):
- Brain Imaging Centre, HUN-REN Centre for Natural Sciences, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
The HUN-MLI-BRAIN Steering Committee and Management Group are open to requests from external researchers for data collected in this study. Applicants will be asked to submit a study protocol, including the research question, planned analysis, and data required. The Committees will evaluate this plan (i.e., relevance of the research question, suitability of data, quality of proposed analyses, planned/ongoing HUN-MLI-BRAIN analyses, and other matters) on a case-by-case basis and provide the data or reject the request. Shared data will encompass the data dictionary and de-identified data only. Any analysis will be conducted in collaboration with the HUN-MLI-BRAIN Management Group. Access is subject to the HUN-MLI-BRAIN legal framework. An access agreement will be prepared and signed by both parties.
Supporting Information: Study Protocol
Time Frame: The trial Steering Committee and Management Group will consider applications for data after the trials results have been published and data will be made available according to the terms of the access agreement.
Access Criteria: As described above in the Plan Description.

REFERENCES:
- [Background] Barbera M, Lehtisalo J, Perera D, Aspo M, Cross M, De Jager Loots CA, Falaschetti E, Friel N, Luchsinger JA, Gavelin HM, Peltonen M, Price G, Neely AS, Thunborg C, Tuomilehto J, Mangialasche F, Middleton L, Ngandu T, Solomon A, Kivipelto M; MET-FINGER study team. A multimodal precision-prevention approach combining lifestyle intervention with metformin repurposing to prevent cognitive impairment and disability: the MET-FINGER randomised controlled trial protocol. Alzheimers Res Ther. 2024 Jan 31;16(1):23. doi: 10.1186/s13195-023-01355-x. PMID 38297399
- [Background] Barbera M, Perera D, Matton A, Mangialasche F, Rosenberg A, Middleton L, Ngandu T, Solomon A, Kivipelto M. Multimodal Precision Prevention - A New Direction in Alzheimer's Disease. J Prev Alzheimers Dis. 2023;10(4):718-728. doi: 10.14283/jpad.2023.114. PMID 37874092